CLINICAL TRIAL: NCT07300969
Title: A Phase 2 Double-blind, Randomised, Placebo-controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of DT-101 in Adults With Major Depressive Disorder (MDD)
Brief Title: A Study to Evaluate the Effectiveness of DT-101 in Patients With Depression
Acronym: Tarian-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Draig Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DT-101/201
Record Dates: First submitted 2025-12-22; First posted 2025-12-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: MDD; Depression; DT-101; randomized; placebo controlled; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DT-101 A (Experimental)
  Interventions: Drug: DT-101
- DT-101 B (Experimental)
  Interventions: Drug: DT-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DT-101 — DT-101 A
  Arms: DT-101 A
Drug: DT-101 — DT-101 B
  Arms: DT-101 B
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if DT-101 can treat depression in adults. The effect of DT-101 will be compared to placebo. Subjects will attend the clinic every couple of weeks complete general health checks and complete questionnaires.

DETAILED DESCRIPTION:
The purpose of this study is to compare DT-101 and placebo in adult participants with MDD. The study will also evaluate how safe and well tolerated the study drug is. The clinical study staff will check participants' suitability to take part in the clinical research study by performing physical and neurological examinations, obtaining blood and urine samples, conducting clinical assessments and reviewing medical and treatment history. These tests and assessments will continue throughout the study with the purpose of checking the participants' ongoing suitability and to collect data to analyze the effect that DT-101 may have on their depression symptoms. Participants will also have blood samples taken to allow analysis of how DT-101 is absorbed and used by the body (PK sampling), some blood samples may be retained in order to perform future research that may be useful when looking at whether genetics affects how a person responds to DT-101 (PGx sampling)

ELIGIBILITY:
Inclusion Criteria:

* The participant is able to read, understand and communicate in the local language used at the study site, and is willing to provide written informed consent
* Male or female (assigned at birth, inclusive of all gender identities) participant must be 18 to 75 years of age, inclusive at the time of signing the informed consent.
* Has recurrent depression (defined as at least one prior episode excluding the current one), as diagnosed by DSM 5-TR (Diagnostic and Statistical Manual of Mental Disorders, 2022).

Exclusion Criteria:

* Pregnant or breastfeeding or plans to become pregnant during the study.
* Unstable medical condition or unstable chronic disease.
* Significant neurological abnormality.
* History of moderate or severe alcohol or drug use disorder as per DSM-5-TR in the 6 months prior to Screening.
* History of seizure.
* In the investigator's opinion, the participant is not capable of adhering to the protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total Montgomery Åsberg depression rating scale (MADRS) score, at Day 42 | from enrollment to day 42

SECONDARY OUTCOMES:
Change from baseline in Clinician Global Impression of severity (CGI-S), at Day 42 | From enrollment until day 42

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Draig Clinical Site, Bentonville, Arkansas
  - Draig Clinical Site, Little Rock, Arkansas
  - Draig Clinical Site, Oceanside, California
  - Draig Clinical Site, San Diego, California
  - Draig Clinical Site, Torrance, California
  - Draig Clinical Site, Miami, Florida
  - Draig Clinical Site, New Port Richey, Florida
  - Draig Clinical Site, Atlanta, Georgia
  - Draig Clinical Site, Decatur, Georgia
  - Draig Clinical Site, Gaithersburg, Maryland
  - Draig Clinical Site, Las Vegas, Nevada
  - Draig Clinical Site, Marlton, New Jersey
  - Draig Clinical Site, Media, Pennsylvania
  - Draig Clinical Site, Austin, Texas
  - Draig Clinical Site, Richardson, Texas
  - Draig Clinical Site, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No